CLINICAL TRIAL: NCT05805137
Title: Monitoring of Venous Ulcers Using a Bioimpedance Measurement Based Method and System
Acronym: WoundWatch®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CutoSense Oy (Industry)
Collaborators: University Clinical Centre, Gdansk (Other); Medical University of Gdansk (Other); Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WW001; R23094L (WW001 TAYS) (Registry Identifier: Tampere University Hospital)
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Venous Ulcer
Keywords: Venous ulcer; Monitoring; Bioimpedance; Electrode array; Wound dressing
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study subject with venous ulcer (Experimental): The subjects will be monitored using the WoundWatch wound management system two to three study visits per week until the venous ulcer has healed (surface area has decreased at least 90%) or up to two months.
  Interventions: Device: WoundWatch® wound monitoring system

INTERVENTIONS:
Device: WoundWatch® wound monitoring system — eDressing will be applied along with the compression therapy and the standard absorbing dressings. The subjects will be monitored using the WoundWatch® system. The subjects will have two to three study visits per week until the venous ulcer has healed (surface area has decreased at least 90%) or up to two months.
  Other Names: Bioimpedance measurement of wound healing

SUMMARY:
The purpose of this study is to investigate the functionality of a new type of wound monitoring method and measurement system for monitoring healing of venous ulcers. The system is consisted of a wound dressing with electrodes (eDressing), a bioimpedance measurement device and a mobile phone application.

DETAILED DESCRIPTION:
The technical principle of the monitoring method is based on the quasimonopolar bioimpedance measurement. The measurement system consists of a bioimpedance measuring device, a wound dressing with electrodes (eDressing) and a mobile application for use with a mobile phone.

The electrode dressing is placed on top of a wound, in contact with the wound tissue. The other necessary dressing layers (such as absorbent dressings and compression bandages) are placed over the electrode dressing. The electrode dressing is kept on the wound for maximum of seven consecutive days. The electrode dressing can be removed and replaced when needed due to medical reasons. Other dressings can be changed considered necessary.

During a study subject visit, the bioimpedance measurement is made using the device, the uppermost dressings are opened carefully and it is ensured that the wound condition is as expected. Upon the replacement of the electrode dressing, the wound is photographed and documented. The wound area is measured, and the findings are recorded.

A maximum of 20 subjects with venous ulcers will be recruited for the study in two study sites (Gdansk, Poland and Tampere, Finland).

Adult subjects (≥18 years) with venous ulcer who are applicable for compression therapy treatment, whose ulcer is not wider than 5 cm and does not excrete excessively can be recruited to the study. Previous surgical venous procedure is not an exclusion criterion for enrollment, but surgical procedure can not be performed during the study.

A subject shall visit the clinic 2-3 times a week, according to the doctor's or study nurse's assessment. Wound healing is monitored until the wound re-epithelized (>90% of initial wound surface area) or maximum two months. Thus, there will be a maximum of 24 study visits per subject.

In addition to scientific objectives, the results of this study are also used as part of clinical evidence when submitting the technical documentation to Notified Body for assessment of the conformity of the device before being placed on the market.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* The subject has a chronic lower extremity ulcer with a primary etiology of venous insufficiency. The previous venous procedure is not an obstacle to the study
* Compression therapy can be implemented
* The wound is not wider than 5 cm and the electrode dressing can be placed on the wound as intended. The wound should be located above the ankle, on the skin area where the electrode dressing can be placed properly.
* The wound is not deep with steep edges or cavity-like
* The wound is not highly excreting
* The wound can be expected to heal within two months (area reduced ≥ 90% from baseline)
* The subject gives consent to the study and commits to following the instructions of the medical staff

Exclusion Criteria:

* Clinical wound infection at the time of the study
* The subject has an intravenous (in Tampere: A venous operation) procedure within 2 months
* Significant arterial circulatory disorder or adherence problem that prevents compression therapy (in Tampere: Contraindication for compression therapy, e.g. significant arterial circulatory disorder or severe heart failure)
* Subject movement 2-3 times a week during the study to the study site is difficult to arrange (in Tampere: Subject not able to commit to study visits 2-3 times a week.)
* Diagnosed epoxy resin allergy
* Any other reasons of potential study subject non-compliance by the opinion of the investigator

Additional local exclusion criteria in Tampere site:

* Special groups, such as pregnant women/patients trying to conceive during the study or patients with reduced autonomy
* Subject with any implantable electrical device. Such as pacemaker or implanted defibrillator. Patient has other electrically conductive implanted material in legs. Such as a metallic prostheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Wound Status Index (WSI) vs. wound surface area | From admission to discharge, up to 8 weeks.
  Correlation analysis between the WSI and the wound surface area.
Wound Status Index (WSI) vs. wound surface area | From admission to discharge, up to 8 weeks.
  Bland-Altman (agreement) analysis between the WSI and the wound surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Spychalski, MD, Ph.D., Principal Investigator — Department of General, Endocrine and Transplant Surgery, Medical University of Gdansk
Locations (2):
- TAYS Haavakeskuksen poliklinikka, Tampere, Finland
- University Clinical Centre, Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kekonen A, Bergelin M, Eriksson JE, Vaalasti A, Ylanen H, Kielosto S, Viik J. Bioimpedance method for monitoring venous ulcers: Clinical proof-of-concept study. Biosens Bioelectron. 2021 Apr 15;178:112974. doi: 10.1016/j.bios.2021.112974. Epub 2021 Jan 7. PMID 33524705
- [Background] Kekonen A, Bergelin M, Johansson M, Kumar Joon N, Bobacka J, Viik J. Bioimpedance Sensor Array for Long-Term Monitoring of Wound Healing from Beneath the Primary Dressings and Controlled Formation of H2O2 Using Low-Intensity Direct Current. Sensors (Basel). 2019 May 31;19(11):2505. doi: 10.3390/s19112505. PMID 31159298
- [Background] Kekonen A, Bergelin M, Eriksson JE, Vaalasti A, Ylanen H, Viik J. Bioimpedance measurement based evaluation of wound healing. Physiol Meas. 2017 Jun 22;38(7):1373-1383. doi: 10.1088/1361-6579/aa63d6. PMID 28248191
- [Background] Antoszewska M, Spychalski P, Kekonen A, Viik J, Baranska-Rybak W. Bioimpedance sensor array for monitoring chronic wounds: Validation of method feasibility. Int Wound J. 2024 Aug;21(8):e14899. doi: 10.1111/iwj.14899. PMID 39099180
- See also: CutoSense Oy homepage (Sponsor) — https://cutosense.fi/